CLINICAL TRIAL: NCT03786172
Title: Smoking Cessation Intervention for Head and Neck Cancer Patients: A Prospective Randomised Controlled Trial
Brief Title: Efficacy of Smoking Cessation Intervention for Head and Neck Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint-Joseph University (Other)
Collaborators: Hotel Dieu de France Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEHDF600
Record Dates: First submitted 2015-12-10; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Smoking; Head and Neck Neoplasms
Keywords: Smoking cessation; Intervention; Head and Neck neoplasms; Cognitive therapy
MeSH Terms: conditions — Smoking; Head and Neck Neoplasms; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoking cessation Intervention (Experimental): Standardised counseling session + motivational gadget + Nicotine replacement therapy (NRT)
  Interventions: Behavioral: Smoking cessation Intervention
- Usual care (Active Comparator): A 10-second brief advice to quit smoking
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Smoking cessation Intervention — * A 10 to 15 minute standardised counseling session performed peri-operatively by an ENT resident, and based on the 5 "A"s motivational interviewing model (Ask, Advise, Assess, Assist, Arrange)
  * A motivational gadget distributed to the patients
  * Nicotine replacement therapy (NRT), consisting of nicotine transdermal patches for 8 weeks, offered to the patients
  Arms: Smoking cessation Intervention
Behavioral: Usual care — A 10-second brief advice to quit smoking, performed peri-operatively by an ENT resident
  Arms: Usual care

SUMMARY:
The purpose of this study is to determine whether a brief smoking ENT-resident-based intervention increased smoking cessation in patients with Head and Neck cancer attending a Lebanese university hospital, as compared with usual care.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the effectiveness of a brief smoking physician-based intervention on smoking-cessation rates in Head and Neck cancer adult patients. The secondary objective is to assess predictors of long-term smoking cessation in such patients.

After an initial assessment of demographic, clinical and smoking characteristics, the patients are randomised (based on a computer randomisation program) in 2 groups:

* Group 1 will receive the usual care in Lebanon, which consists of a brief advice to quit (10 seconds)
* Group 2 will receive a brief (10-15 minutes) standardised smoking cessation counseling session peri-operatively (immediately before or after surgery), by an ENT residents, based on the 5 "A"'s motivational interviewing model:
* Ask (screen for tobacco use)
* Advise (provide a personalised and strong quit message)
* Assess (evaluate the smoker's willingness and readiness to quit)
* Assist (provide cessation counseling, pharmacotherapy, self-help guides)
* Arrange (for followup to prevent relapse, and evaluate cessation progress) A motivational gadget will be distributed to group 2 patients. They will also be offered nicotine replacement therapy (nicotine transdermal patches) for a total of 8 weeks. This will be followed by a telephone boost session after 6 weeks.

The follow-up at 3, 6 and 12 months will be done, for the 2 groups, by a person not implicated in either the randomisation or the intervention (single-blind), in person or, if impossible, by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Head and Neck cancer
* Patients hospitalised from biopsy or surgery
* Current smokers = smokers in the past 3 months
* Reachable by phone

Exclusion Criteria:

* Nonsmokers in the past 3 months
* Current drug dependance
* Pregnant women
* Psychiatric conditions
* Patients under current smoking cessation intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence abstinence | 12 months
  The patient is considered abstinent if he reported not smoking for at least 7 days before the interview

SECONDARY OUTCOMES:
continuous abstinence | 12 months
  continuous abstinence from smoking at the time of follow-up, since the quit date

CONTACTS AND LOCATIONS:
Overall Officials: Amine Haddad, MD ENT, Study Director — Hotel Dieu de France Hospital
Locations (2):
- Lebanon (2):
  - Saint-Joseph university, Beirut
  - Hôtel-Dieu De France University Hospital, Beirut

REFERENCES:
- [Background] 2008 PHS Guideline Update Panel, Liaisons, and Staff. Treating tobacco use and dependence: 2008 update U.S. Public Health Service Clinical Practice Guideline executive summary. Respir Care. 2008 Sep;53(9):1217-22. No abstract available. PMID 18807274
- [Background] Nayan S, Gupta MK, Strychowsky JE, Sommer DD. Smoking cessation interventions and cessation rates in the oncology population: an updated systematic review and meta-analysis. Otolaryngol Head Neck Surg. 2013 Aug;149(2):200-11. doi: 10.1177/0194599813490886. Epub 2013 May 28. PMID 23715685
- [Background] Duffy SA, Ronis DL, Valenstein M, Lambert MT, Fowler KE, Gregory L, Bishop C, Myers LL, Blow FC, Terrell JE. A tailored smoking, alcohol, and depression intervention for head and neck cancer patients. Cancer Epidemiol Biomarkers Prev. 2006 Nov;15(11):2203-8. doi: 10.1158/1055-9965.EPI-05-0880. PMID 17119047
- [Background] Schnoll RA, Rothman RL, Wielt DB, Lerman C, Pedri H, Wang H, Babb J, Miller SM, Movsas B, Sherman E, Ridge JA, Unger M, Langer C, Goldberg M, Scott W, Cheng J. A randomized pilot study of cognitive-behavioral therapy versus basic health education for smoking cessation among cancer patients. Ann Behav Med. 2005 Aug;30(1):1-11. doi: 10.1207/s15324796abm3001_1. PMID 16097900
- [Background] Schnoll RA, Zhang B, Rue M, Krook JE, Spears WT, Marcus AC, Engstrom PF. Brief physician-initiated quit-smoking strategies for clinical oncology settings: a trial coordinated by the Eastern Cooperative Oncology Group. J Clin Oncol. 2003 Jan 15;21(2):355-65. doi: 10.1200/JCO.2003.04.122. PMID 12525530
- [Background] Rigotti NA, Munafo MR, Stead LF. Interventions for smoking cessation in hospitalised patients. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD001837. doi: 10.1002/14651858.CD001837.pub2. PMID 17636688
- [Background] Wakefield M, Olver I, Whitford H, Rosenfeld E. Motivational interviewing as a smoking cessation intervention for patients with cancer: randomized controlled trial. Nurs Res. 2004 Nov-Dec;53(6):396-405. doi: 10.1097/00006199-200411000-00008. PMID 15586136
- [Background] Gosselin MH, Mahoney MC, Cummings KM, Loree TR, Sullivan M, King BA, Warren G, Hyland A. Evaluation of an intervention to enhance the delivery of smoking cessation services to patients with cancer. J Cancer Educ. 2011 Sep;26(3):577-82. doi: 10.1007/s13187-011-0221-3. PMID 21503842
- [Background] Schnoll RA, Rothman RL, Newman H, Lerman C, Miller SM, Movsas B, Sherman E, Ridge JA, Unger M, Langer C, Goldberg M, Scott W, Cheng J. Characteristics of cancer patients entering a smoking cessation program and correlates of quit motivation: implications for the development of tobacco control programs for cancer patients. Psychooncology. 2004 May;13(5):346-58. doi: 10.1002/pon.756. PMID 15133775
- [Background] Gorin SS, Heck JE. Meta-analysis of the efficacy of tobacco counseling by health care providers. Cancer Epidemiol Biomarkers Prev. 2004 Dec;13(12):2012-22. PMID 15598756
- [Background] Sharp L, Johansson H, Fagerstrom K, Rutqvist LE. Smoking cessation among patients with head and neck cancer: cancer as a 'teachable moment'. Eur J Cancer Care (Engl). 2008 Mar;17(2):114-9. doi: 10.1111/j.1365-2354.2007.00815.x. PMID 18302647
- [Background] Gritz ER, Carr CR, Rapkin D, Abemayor E, Chang LJ, Wong WK, Belin TR, Calcaterra T, Robbins KT, Chonkich G, et al. Predictors of long-term smoking cessation in head and neck cancer patients. Cancer Epidemiol Biomarkers Prev. 1993 May-Jun;2(3):261-70. PMID 8318879